CLINICAL TRIAL: NCT06988475
Title: DETERMINE (Determining Extended Therapeutic Indications for Existing Drugs in Rare Molecularly Defined Indications Using a National Evaluation Platform Trial): An Umbrella-Basket Platform Trial to Evaluate the Efficacy of Targeted Therapies in Rare Adult, Paediatric and Teenage/Young Adult (TYA) Cancers With Actionable Genomic Alterations, Including Common Cancers With Rare Actionable Alterations. Treatment Arm 06: Capmatinib in Adult Patients With Cancers Harbouring MET Dysregulations
Brief Title: DETERMINE Trial Treatment Arm 06: Capmatinib in Adult Patients With Cancers Harbouring MET Dysregulations
Acronym: DETERMINE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: University of Birmingham (Other); Royal Marsden NHS Foundation Trust (Other); Novartis Pharmaceuticals (Industry); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/21/004 - Treatment Arm 6
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumour; Haematological Malignancy; Malignant Neoplasm; Neoplasms by Histologic Type; Neoplasms by Site; Cancer; Malignancy; Glioma; Neuroblastoma; Gastric Cancer; Soft Tissue Sarcoma
Keywords: adult; capmatinib; MET Tyrosine Kinase Receptor; MET exon 14 skipping; MET amplifications; MET fusions; MET activating mutations; MET dysregulations; Antineoplastic Agents; cancer; malignancy; Malignant Neoplasms; Molecular Targeted Therapy; Mutation; Neoplasms by Histologic Type; Neoplasms by Site; Precision Medicine; Protein Kinase Inhibitors; Rare; Tumour-agnostic; METex14 skipping
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms; Neoplasms by Histologic Type; Neoplasms by Site; Glioma; Neuroblastoma; Stomach Neoplasms; Sarcoma | interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm 06: Capmatinib (Experimental): This capmatinib treatment arm is for adult partients with cancers harbouring MET dysregulations.
  Interventions: Drug: Capmatinib

INTERVENTIONS:
Drug: Capmatinib — Patients will be administered capmatinib orally at a daily dose of 800 mg consisting of 400 mg (two 200mg tablets) twice daily. Each cycle of treatment will consist of 28 days and patients may continue on treatment until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.

SUMMARY:
This clinical trial is looking at a drug called capmatinib. Capmatinib is approved as standard of care treatment for adult patients with certain types of lung cancer. This means it has gone through clinical trials and been approved by the Medicines and Healthcare products Regulatory Agency (MHRA) in the UK.

Capmatinib works in patients with lung cancer with a particular mutation in their cancer known as a METex14 skipping mutation.

Investigators now wish to find out if it will be useful in treating patients with other cancer types which have the same mutation or other specific mutations or changes which take place in the MET gene. If the results are positive, the study team will work with the NHS and the Cancer Drugs Fund to see if these drugs can be routinely accessed for patients in the future.

This trial is part of a trial programme called DETERMINE. The programme will also look at other anti-cancer drugs in the same way, through matching the drug to rare cancer types or ones with specific mutations.

DETAILED DESCRIPTION:
DETERMINE Treatment Arm 06 (capmatinib) aims to evaluate the efficacy of capmatinib in adult patients with rare* cancers harbouring MET dysregulations and in common cancers where MET dysregulations are considered to be infrequent.

*Rare is defined generally as incidence less than 6 cases in 100,000 patients (includes paediatric and teenagers/young adult cancers) or common cancers with rare alterations.

This treatment arm has a target sample size of 30 evaluable patients. Sub-cohorts may be defined and further expanded to a target of 30 evaluable patients each.

The ultimate aim is to translate positive clinical findings to the NHS (Cancer Drugs Fund) to provide new treatment options for rare adult cancers.

OUTLINE:

Pre-screening: The Molecular Tumour Board makes a treatment recommendation for the patient based on molecularly-defined cohorts (See information on Master Screening Protocol below).

Screening: Consenting patients undergo biopsy and collection of blood samples for research purposes.

Treatment: Patients will receive capmatinib until disease progression without clinical benefit, unacceptable adverse events (AEs) or withdrawal of consent. Patients will also undergo collection of blood samples at various intervals while receiving treatment and at End of Treatment (EoT).

After completion of study treatment, patients are followed up every 3 months for 2 years.

THE DETERMINE TRIAL MASTER (SCREENING) PROTOCOL:

Please see DETERMINE Trial Master (Screening) Protocol record (NCT05722886) for information on the DETERMINE Trial Master Protocol and applicable documents.

ELIGIBILITY:
THE PATIENT MUST FULFIL THE ELIGIBILITY CRITERIA WITHIN THE DETERMINE MASTER PROTOCOL (NCT05722886) AND WITHIN THE TREATMENT ARM 06 (CAPMATINIB) OUTLINED BELOW*

*When capmatinib-specific inclusion/exclusion criteria or precautions below differ from those specified in the Master Protocol, the capmatinib-specific criteria will take precedence.

Inclusion criteria:

A. Confirmed diagnosis of a MET-positive malignancy using an analytically next-generation sequencing method (METex14 skipping, MET amplification, MET fusion, or MET activating mutation).

B. Adult patients ≥18 years old.

C. Women of childbearing potential are eligible, provided that they meet the following criteria:

* Have a negative serum or urine pregnancy test before enrolment, and
* Agree to use one form of highly effective birth control method (a method that can achieve a failure rate of <1% when used consistently and correctly), such as:

I. combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation [oral, intravaginal or transdermal])

II. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable)

III. intrauterine device (IUD)

IV. Intrauterine hormone-releasing system (IUS)

V. bilateral tubal occlusion

VI. vasectomised partner

VII. sexual abstinence

Effective from the first administration of capmatinib, throughout the trial and for seven days after the last administration of capmatinib.

D. Male patients with partners who are women of childbearing potential are eligible provided that they agree to the following, from first administration of capmatinib, throughout the trial and for seven days after the last administration of capmatinib:

* Agree to take measures not to father children by using a barrier method of contraception (e.g. condom) or sexual abstinence.
* Non-vasectomised male patients with partners who are women of childbearing potential must also be willing to ensure that their partner uses a highly effective method of contraception, as in criterion C above.
* Male patients with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom) to prevent drug exposure of the foetus or neonate.

All male patients must refrain from donating sperm for the same period.

E. Patients must be able and willing to undergo a fresh biopsy at baseline and blood samples for translational research. Note that for patients with haematological malignancies or neuroblastomas, blood, bone marrow aspiration and/or trephine or lymph node biopsy samples may be taken.

F. Adequate organ function as per haematological and biochemical indices within the ranges defined in the protocol. These measurements should be performed to confirm the patient's eligibility.

Exclusion criteria:

A. Diagnosis of NSCLC with METex14 skipping mutation or MET amplification.

B. Prior treatment with a selective MET inhibitor or HGF-targeting therapy unless genetic profile demonstrates a mechanism of resistance known to be potentially sensitive to capmatinib.

C. Carcinomatous meningitis.

D. Presence or history of additional malignant disease that has been diagnosed and/or required therapy within the past three years. Exceptions to this exclusion include: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.

E. Presence or history of interstitial lung disease (ILD) and/or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention) and evidence of active pneumonitis on screening chest computed tomography (CT) scan. Prior localised radiotherapy related pneumonitis is permitted if resolved and off steroids and asymptomatic for at least six months.

F. Clinically significant, uncontrolled heart disease such as:

* Unstable angina within three months prior to screening
* Myocardial infarction within three months prior to screening
* History of documented congestive heart failure (New York Heart Association functional classification III-IV)
* Uncontrolled hypertension defined by a systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg, with or without antihypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening.

Patients with a cerebrovascular event (including stroke or transient ischaemic attack [TIA]) within three months before screening.

• Patients with primary CNS tumours may be considered unless intra-tumoural bleeding has occurred within two weeks of the first dose of capmatinib, and patients with punctate CNS haemorrhages <3 mm may be considered.

G. History or current diagnosis of electrocardiogram (ECG) abnormalities indicating significant risk of safety for patients participating in the trial such as:

* Concomitant clinically significant cardiac arrhythmias (atrial and ventricular), e.g., sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker
* History of familial long QT syndrome or known family history of Torsades de Pointes
* Resting QTcF (Corrected QT interval by Fridericia formula) ≥450 msec (male) or ≥460 msec (female) at screening ECG (as a mean of triplicate ECG)

H. Major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within four weeks prior to starting trial treatment (two weeks for resection of brain lesions) or patients who have not recovered from side effects of such procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and patients can be enrolled in the trial at least one week after the procedure.

I. Patients receiving treatment with strong inducers of cytochrome P450 (CYP) 3A that cannot be discontinued at least one week prior to the start of treatment with capmatinib and for the duration of the trial.

J. Any clinically significant concomitant disease or condition (or its treatment) that could interfere with the conduct of the trial (including absorption of oral medications) that would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this trial.

K. Any impairment of gastrointestinal (GI) function or GI disease that may significantly alter the administration or absorption of capmatinib (e.g., Crohn's disease, ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome or short gut syndrome). Unable to swallow capmatinib intact, without chewing or crushing the tablets (as per the dosing schedule).

L. Active infections including, but not limited to, hepatitis B virus (HBV), hepatitis C virus (HCV) and human immunodeficiency virus (HIV). Screening for known chronic conditions is not required. Patients with known serological evidence of chronic HBV or HCV infection whose disease is controlled under antiviral therapy according to local regulation are eligible. Patients with history of testing positive for human immunodeficiency virus (HIV) infection are eligible provided the each of the following conditions are met:

* CD4 count ≥350/μL;
* undetectable viral load;
* receiving antiretroviral therapy (ART) that does not interact with IMP (patients should be on established ART for at least four weeks); and
* no HIV/ acquired immune deficiency syndrome-associated opportunistic infection in the last 12 months.

M. Known hypersensitivity to any of the excipients of capmatinib.

N. Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the two weeks prior to trial entry to manage CNS symptoms. Primary brain or CNS malignancies are allowed providing the patient is clinically stable (if corticosteroids are required, they must be at a stable or decreasing dose for at least 14 days prior to Cycle 1 Day 1). If patients are on corticosteroids for endocrine deficiencies or tumour-associated symptoms other than CNS related, the dose must have been stabilised (or decreasing) for at least five days before Cycle 1 Day 1.

O. Patients receiving treatment with any enzyme-inducing anticonvulsant that cannot be discontinued at least one week before first dose of capmatinib, and for the duration of the trial. Patients on non-enzyme-inducing anticonvulsants are eligible.

P. Female patients who are pregnant, breastfeeding or planning to become pregnant during the trial or for seven days following their last dose of capmatinib.

Q. Patients who were administered a live, attenuated vaccine within 28 days prior to enrolment, or anticipation of need for such a vaccine during capmatinib treatment or within six months after the final dose of capmatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) | Disease assessments to be performed up to 24 weeks from the start of trial treatment.
  OR is defined as the confirmed occurrence of either a Complete Response (CR) or Partial Response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 criteria (or immune related [ir]-RECIST or standard imaging criteria for specific disease e.g. Response Evaluation in Neuro Oncology criteria [RANO]). In patients with leukaemia, OR will be defined as the occurrence of CR, CRi (CR incomplete neutrophil recovery) or CRp (CR with incomplete platelet recovery). The trial will report the proportion of patients with an OR and 95% credible interval.
Durable Clinical Benefit (DCB) | Disease assessments to be performed up to 24 weeks from the start of trial treatment.
  DCB is defined as the absence of disease progression for at least 24 weeks from the start of trial treatment according to RECIST Version 1.1 criteria (or ir-RECIST or standard imaging criteria for specific disease e.g. RANO criteria) and, where relevant (e.g. for haematological malignancies), by standard bone marrow response assessment criteria. Alternative definitions of DCB based on different time points may be pre-specified for particular sub-cohorts if 24 weeks is not clinically relevant. The trial will report the proportion of patients with a DCB and 95% credible interval.

SECONDARY OUTCOMES:
Duration of response (DR) | Disease assessment performed every 2 cycles of capmatinib (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of capmatinib for up to 2 years.
  DR is defined as the time from the date of the first confirmed CR or PR according to RECIST 1.1 or ir-RECIST or standard imaging criteria for specific disease (e.g. RANO criteria) to the date of disease progression. The trial will report the median DR and 95% credible interval.
Best percentage change in sum of target lesion / index lesion diameters (PCSD) | Disease assessment performed every 2 cycles of capmatinib (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of capmatinib for up to 2 years.
  PCSD is defined as the greatest decrease or least increase in the sum of target lesion diameters (RECIST) or index lesion diameters (irRECIST) as a percentage compared to the baseline measurement. The trial will report the mean PCSD and 95% credible interval.
Time to treatment discontinuation (TTD) | From first dose of capmatinib to discontinuation of trial treatment up to 5 years with an average calculated and presented with results entry.
  TTD is defined as the time from date of starting trial treatment to date of discontinuing trial treatment, in days estimated by the median of the posterior inverse gamma probability distribution. The trial will report the median TTD and 95% credible interval.
Progression-Free Survival time (PFS) | Disease assessment performed every 2 cycles of capmatinib (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of capmatinib for up to 2 years.
  PFS is defined as the time from date of starting trial treatment to date of progression or date of death without a previous progression recorded estimated by the median of the posterior inverse gamma probability distribution.
Time to Progression (TTP) | Disease assessment performed every 2 cycles of capmatinib (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of capmatinib for up to 2 years.
  TTP is defined as the time from date of starting trial treatment to date of progression or date of death without recorded progression censored rather than events. The trial will report the median TTP and 95% credible interval.
Growth Modulation Index (GMI) | Disease assessment performed every 2 cycles of capmatinib (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of capmatinib for up to 2 years.
  GMI is defined as the ratio of TTP with the trial protocol treatment to TTP on the most recent prior line of therapy. The trial will report the mean GMI and 95% credible interval.
Overall Survival time (OS) | Time of death or up to 2 years after the EoT visit.
  OS is defined as the time from date of starting trial treatment to date of death from any cause estimated by the median of the posterior normal probability distribution.
Occurrence of at least one Suspected Unexpected Serious Adverse Reaction (SUSAR) | From the time of consent until 28 days after last dose of capmatinib (up to 5 years) or until patient starts another anti-cancer therapy, whichever came first. An average time frame will be presented with results entry.
  The trial will report the number of patients who experience at least one SUSAR to capmatinib.
Occurrence of at least one Grade 3, 4 or 5 capmatinib related AE | From the time of consent until 28 days after last dose of capmatinib (up to 5 years) or until patient starts another anti-cancer therapy, whichever came first. An average time frame will be presented with results entry.
  Number of patients who experience at least one capmatinib related Grade 3, 4 or 5 AE according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0
EORTC-QLQ-30-Standardised Area Under Summary Score Curve (QLQSAUC) | QoL surveys performed at baseline every cycle (every cycle is 28 days) and after interrupting treatment (up to 5 years).
  Multiple measures of Quality of Life (QoL) will be generated from patient completion of the European Organisation for Research and Treatment of Cancer QLQC30 (EORTC-QLQ-C30) questionnaire (15 measures). For each patient the Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean QLQSAUC and 95% credible interval.
EQ-5D Standardised Area Under Index Value Curve (EQ5DSAUC) | QoL surveys performed prior to inclusion, every cycle (each cycle is 28 days) and at EoT visit (up to 5 years).
  Two measures of QoL will be generated from patient completion of the EQ-5D-5L questionnaire. For each measure, scores based on responses from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean EQ5DSAUC and 95% credible interval.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Krebs, Dr, Principal Investigator — The Christie Hospital
Locations (17):
- United Kingdom (17):
  - Belfast City Hospital, Belfast
  - University Hospital Birmingham, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - The Beatson Hospital, Glasgow
  - Leicester Royal Infirmary, Leicester
  - University College London Hospital, London
  - Guy's Hospital, London
  - The Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Freeman Hospital, Newcastle
  - Churchill Hospital, Oxford
  - Western Park Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified patient data will be shared with researchers whose proposed use of the data is approved by a review committee of the Sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All requests for data relating to this treatment arm that are made within 5 years from last patient last visit for the capmatinib treatment arm will be considered; requests made subsequently will be considered where possible.
Access Criteria: When a request has been approved, Cancer Research UK will provide access to the de-identified individual patient-level data and appropriate supporting information. A signed Data Sharing Agreement must be in place before accessing requested information. Requests should be submitted to drugdev@cancer.org.uk.

REFERENCES:
- See also: Overview of the DETERMINE trial — http://CRUK.org/determine
- See also: ClinicalTrials.gov record for DETERMINE Trial Master Screening Protocol (NCT05722886). — https://clinicaltrials.gov/ct2/show/NCT05722886